CLINICAL TRIAL: NCT05130554
Title: XEN45 in the Treatment of Chinese Patients With Primary Open-angle Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021KYPJ172
Record Dates: First submitted 2021-11-06; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Glaucoma; Glaucoma, Open-Angle; Surgery
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XEN45 (Experimental): The effect of XEN45 surgery on patients with primary open-angle glaucoma
  Interventions: Procedure: XEN45 gel stent implantation

INTERVENTIONS:
Procedure: XEN45 gel stent implantation — The XEN45 gel implant is a collagen tube with a length of 6 mm and a diameter of 45 µm, which creates a new channel for drainage of aqueous humor by connecting the anterior chamber and the subconjunctival space. The implant is composed of porcine gelatin cross-linked with glutaraldehyde, and has good biocompatibility and tolerance.This treatment method has excellent safety and effectiveness in reducing the intraocular pressure of patients with open-angle glaucoma. At the same time, the operation is simple and safe.
  Other Names: XEN

SUMMARY:
Glaucoma is the second most common blindness disease in the world, second only to cataracts. The current treatment of glaucoma is mainly to reduce intraocular pressure.At present, two commonly used surgical methods are trabeculectomy and implantation of drainage valve. These methods are superior to drug treatment in reducing intraocular pressure, but the effect duration of these two methods is not long, and there may be serious complications and failure.

Compared with traditional glaucoma surgery, MIGS may have better safety.The XEN45 gel implant is a collagen tube with a length of 6 mm and a diameter of 45 µm, which creates a new channel for drainage of aqueous humor by connecting the anterior chamber and the subconjunctival space. The implant is composed of porcine gelatin cross-linked with glutaraldehyde, and has good biocompatibility and tolerance. Therefore, after the advent of XEN45 products, more and more studies have shown that this treatment has excellent safety and effectiveness in reducing intraocular pressure in patients with open-angle glaucoma.

Considering that the XEN45 gel stent has been in the market for a relatively short time, we conducted this prospective study to investigate the effect of XEN45 surgery in the treatment of primary open-angle glaucoma, in order to support ophthalmologists in formulating the best surgical plan for patients. The promotion of this surgical method.

DETAILED DESCRIPTION:
Observation index： The visual acuity, intraocular pressure, slit lamp, ophthalmoscope, traditional vision, UBM and anti-glaucoma drugs before surgery and 1 day, 1 week, 1 month, 3 months, 6 months, and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with POAG;
2. The visual acuity of the affected eye is greater than that of manual operation;
3. Between 18 and 90 years old;
4. No surgery or laser treatment within 90 days;
5. Patients with other types of glaucoma whose intraocular pressure has not been controlled by traditional surgery or medication;
6. The target quadrant has healthy conjunctiva and free movement without scars.

Exclusion Criteria:

1. Angle-closure glaucoma;
2. Active uveitis;
3. Any corneal disease;
4. Patients with eye infections two weeks before the operation;
5. During pregnancy or lactation;
6. Active neovascular glaucoma;
7. Known or suspected allergy or sensitivity to pig products or glutaraldehyde.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-07 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
IOP (intraocular pressure) changes | 3 months after surgery
  Compare the patient's IOP changes before and after surgery. Complete success of the operation was defined as IOP≤21mmhg without any glaucoma drugs. Qualified success is defined as the same intraocular pressure level but with medication. Failure is defined as IOP> 21 mmHg and maximum tolerance of the drug

SECONDARY OUTCOMES:
BCVA（Best corrected vision ability）changes | Baseline (before surgery) and 1 day, 1 week, 1 month, 3 months, 6 months, and 12 months after surgery
  Evaluate the patient's BCVA changes before and after surgery
anti-glaucoma drugs changes | Baseline (before surgery) and 1 day, 1 week, 1 month, 3 months, 6 months, and 12 months after surgery
  Compare the amount of patient's anti-glaucoma drugs before and after surgery
IOP (intraocular pressure) changes | Baseline (before surgery) and 1 day, 1 week, 1 month,6 month and 12 months after surgery
  Compare the patient's IOP changes before and after surgery. Complete success of the operation was defined as IOP≤21mmhg without any glaucoma drugs. Qualified success is defined as the same intraocular pressure level but with medication. Failure is defined as IOP> 21 mmHg and maximum tolerance of the drug

CONTACTS AND LOCATIONS:
Overall Officials: Mingkai Lin, M.D,Ph.D, Study Chair — Zhognshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No